CLINICAL TRIAL: NCT02320045
Title: A Phase 1 Study to Evaluate the Pharmacokinetics of ITCA 650 in Subjects With Mild and Moderate Renal Impairment Compared to the Pharmacokinetics of Subjects With Normal Renal Function
Brief Title: Study to Evaluate Pharmacokinetics of ITCA 650 in Subjects With Renal Impairment Compared to Normal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITCA 650 CLP-109
Record Dates: First submitted 2014-11-26; First posted 2014-12-19 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Normal (Experimental): Normal Subjects estimated creatinine clearance (eGFR) ≥90 mL/min/1.73 m2
  Interventions: Drug: ITCA 650 (Exenatide in osmotic mini pump)
- Group 2: Mild Renal Dysfunction (Experimental): Subjects with Mild Renal Dysfunction estimated creatinine clearance (eGFR) 60-89 mL/min/1.73 m2
  Interventions: Drug: ITCA 650 (Exenatide in osmotic mini pump)
- Goup 3: Moderate Renal Dysfunction (Experimental): Subjects with Moderate Renal Dysfunction estimated creatinine clearance (eGFR) 45-59 mL/min/1.73 m2
  Interventions: Drug: ITCA 650 (Exenatide in osmotic mini pump)
- Group 4: Moderate Renal Dysfunction (Experimental): Subjects with Moderate Renal Dysfunction estimated creatinine clearance (eGFR) >30-44 mL/min/1.73 m2
  Interventions: Drug: ITCA 650 (Exenatide in osmotic mini pump)

INTERVENTIONS:
Drug: ITCA 650 (Exenatide in osmotic mini pump)

SUMMARY:
A Phase 1 study to evaluate the pharmacokinetics of ITCA 650 in subjects with mild and moderate renal impairment compared to the pharmacokinetics of subjects with normal renal function

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 22 and 40 kg/m²
* Subjects meeting pre-defined estimated glomerular filtration rate criteria and creatinine clearance rate

  * Normal (≥90 mL/min/1.73 m2)
  * Mild (60-89 mL/min/1.73 m2)
  * Moderate (45-59 mL/min/1.73 m2)
  * Moderate (>30-44 mL/min/1.73 m2)

Exclusion Criteria:

* History of acute metabolic complications
* Uncontrolled Hypertension
* History of Hypersensitivity to Exenatide
* Cardiovascular Disease
* History of Acute or chronic pancreatitis
* Personal or family history of Multiple endocrine neoplasia type 2
* History of Medullary thyroid cancer
* Severe renal failure, End stage renal disease or dialysis

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
24-h Area under the Curve at steady state (AUCt,ss) | Approximately 67 Days

SECONDARY OUTCOMES:
Rate of adverse events | Approximately 67 Days
Severity of adverse events | Approximately 67 Days
Safety laboratory parameters | Approximately 67 Days
Vital signs | Approximately 67 Days
Electrocardiogram | Approximately 67 Days
Physical exam | Approximately 67 Days

CONTACTS AND LOCATIONS:
Locations (4):
- Intarcia Therapeutics Inc., Boston, Massachusetts, United States
- Germany (3):
  - Study Site, Kiel
  - Study Site, Mannheim
  - Study Site, Mönchengladbach